CLINICAL TRIAL: NCT00618878
Title: The Effects of Electroacupuncture and Laser Therapy on Chronic Neck Pain, A Pilot Study
Brief Title: Electroacupuncture and Laser Therapy on Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: John Zhang, Logan college of chiropractic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD0423070088
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Chronic Neck Pain
MeSH Terms: interventions — Electroacupuncture; Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Electroacupuncture
  Interventions: Procedure: Electroacupuncture
- 2 (Active Comparator): Laser Therapy
  Interventions: Procedure: Laser Therapy

INTERVENTIONS:
Procedure: Electroacupuncture — twice a week for 26 treatments in total
  Other Names: Greatwall Brand KWD-808 I Multi-Purpose Health Device
  Arms: 1
Procedure: Laser Therapy — twice a week for a total of 26 treatments
  Other Names: USA Laser
  Arms: 2

SUMMARY:
The purpose of the study examines the use of electroacupuncture and laser therapy to treat chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* people with chronic neck pain, participants with a VAS level between 3 and 10 will be included in the study

Exclusion Criteria:

* history of cancer, tuberculosis, pacemaker usage, pregnancy, hemophilia, cardiovascular disease, osteoporosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Neck Pain Disability Index Questionnaire, Neck Bournemouth Questionnaire, Revised Oswestry Pain Questionnaire | within 30 days of the last treatment

CONTACTS AND LOCATIONS:
Overall Officials: John Zhang, MD, PhD, Principal Investigator — Logan College of Chiropractic
Locations (1):
- Logan College of Chiropractc, Chesterfield, Missouri, United States